CLINICAL TRIAL: NCT03643900
Title: Clinical Research on the Prophylactic Efficacy of Pancreatic Duct Stenting Combined With Rectal Indomethacin Drug on Post Endoscopic Retrograde Cholangiopancreatography Pancreatitis
Brief Title: The Efficacy of Pancreatic Duct Stenting With Rectal Indomethacin in Preventing Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, chief physician, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018053013
Record Dates: First submitted 2018-06-24; First posted 2018-08-23 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Post-ERCP Pancreatitis; Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indomethacin with stenting group (Experimental): Pancreatic duct stenting and rectal indomethacin 100mg at preoperative 30min in 100 patients
  Interventions: Device: pancreatic duct stenting; Drug: rectal indomethacin
- indomethacin group (Active Comparator): Rectal indomethacin 100mg at preoperative 30min in 100 patients
  Interventions: Drug: rectal indomethacin

INTERVENTIONS:
Device: pancreatic duct stenting — Place the pancreatic duct stent
  Other Names: pancreatic stent
  Arms: indomethacin with stenting group
Drug: rectal indomethacin — rectal indomethacin 100mg at preoperative 30min
  Other Names: Indomethacin Suppositories

SUMMARY:
With the development of endoscopic technology, ERCP has been widely used in the diagnosis and treatment of pancreatobiliary diseases, and has become the first treatment for most of the biliary and pancreatic diseases. Postoperative ERCP pancreatitis (PEP) is the most common and serious complication after ERCP. The purpose of this study was to explore methods for preventing postoperative pancreatitis.

1. Participants: Patients with high-risk factors associated with PEP were included in the no-obvious patients who underwent therapeutic ERCP in our hospital from June 2018 to December 2019.
2. Research methods: Patients were randomly divided into indometacin suppositories, indomethacin suppositories and pancreatic stents.
3. Statistical methods: SPSS 13.0 statistical software was used. The measurement data was expressed as x± s, and t-test or non-parametric test was used. Chi-square test was used for count data.

DETAILED DESCRIPTION:
Patients with high risk factors for PEP who will be examined and diagnosed by ERCP at 2018.06-2019.12 in the First People's Hospital of Hangzhou are randomly divided into two groups.

2. Record the relevant indicators of each group of patients: 1 before and after surgery 3, 12, 24 h serum amylase changes 2 patients with abdominal pain, abdominal distension, fever, vomiting and abdominal signs of change; 3 hospital days; 4 CT severity index (CT severity Index, CTSI score: Balthazar 5 scores were scored as 0 to 4 points; according to the scope of necrosis was divided into no, <33%, 33% to 50%,> 50%, respectively rated as 0, 2, 4 and 6 points. Addition of the two scores is the CTSI score. 5 According to the diagnostic criteria for postoperative ERCP pancreatitis, PEP will be diagnosed in patients with persistent abdominal pain within 24 hours after ERCP and blood amylase increase by more than 3 times the normal value. Observed 2 groups of post-ERCP pancreatitis, severe pancreatitis and adverse events Incidence.

3. Analyze and compare the above indicators and observe the effect of the two methods on the reduction of blood amylase level and incidence of pancreatitis. It is clear that rectal administration of preoperative indomethacin suppository has the same protection against PEP as pancreatic stenting effect.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years old,gender is not limited; Preoperative blood amylase is normal; PEP risk factors during surgery:difficulty in intubation,needle knife incision,intraoperative intubation into the pancreatic duct more than 3 times,the contrast agent in the pancreatic duct is filled; The research procedure is willing to be followed and the informed consent is signed.

Exclusion Criteria:

Myocardial infarction occurred within 3 months; Insufficiency of renal function; Conventional gastrectomy; Preoperative state of shock,such as hypotension(systolic blood pressure less than 90mmHg); Pregnancy and lactation; Allergic to NSAIDs drugs; Partially or completely restricted in the ability to exercise consciousness,without self-determination ability; Are participating in other clinical observation trials or have participated in other clinical trials within 60 days; Cases considered unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
the incidence of PEP | 24 hours
  the rate of patients with PEP

SECONDARY OUTCOMES:
CT severity index | 72 hours
  CT severity Index, CTSI score: Balthazar 5 scores were scored as 0 to 4 points; according to the scope of necrosis was divided into no, <33%, 33% to 50%,> 50%, respectively rated as 0, 2, 4 and 6 points. Addition of the two scores is the CTSI score
the incidence of severe PEP | 7 days
  the rate of patients with severe acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Yang, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No